CLINICAL TRIAL: NCT02002351
Title: Prospective Study on Rehabilitation Patients With Pulmonary Hypertension and Other Pulmonary Diseases
Status: Completed | Type: Observational
Sponsor: Paracelsus Harz Clinic Bad Suderode. (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: ParacelsusHCBS 22/13
Record Dates: First submitted 2013-11-28; First posted 2013-12-05 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2015-01

CONDITIONS: Pulmonary Diseases; Rehabilitation
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary disease

SUMMARY:
This monocentric registry should provide information on the extent how patients with pulmonary diseases such as pulmonary hypertension will benefit from rehabilitation treatment. The data may provide a basis for further prospective studies showing the treatment of patients with pulmonary diseases especially by physical activation.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary Disease

Exclusion Criteria:

* Inability or refusal to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All rehabilitation patients with pulmonary diseases in the Paracelsus-Harz-Clinic Bad Suderode will be included, starting December 2013,ending Novermber 2014.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Data collection | 12 Months
  Characterization of patients with pulmonary hypertension and other pulmonary diseases in a german rehabilitation clinic.

CONTACTS AND LOCATIONS:
Locations (1):
- Paracelsus Harz Clinic Bad Suderode, Quedlinburg, Saxony-Anhalt, Germany